CLINICAL TRIAL: NCT02459522
Title: Bayesian Estimation of Diagnostic Performance of Short-term Heart Rate Variability for Cardiovascular Autonomic Neuropathy Without a Gold Standard
Brief Title: Bayesian Estimation of Diagnostic Performance for Cardiovascular Autonomic Neuropathy
Status: Completed | Type: Observational
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zihui Tang, M.D and Ph.D, Huashan Hospital
Other Study IDs: CANHRVB_Dr.Tang
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Diagnostic Performance of Cardiovascular Autonomic Neuropathy
Keywords: Bayesian estimation; short-term heart rate variability; cardiovascular autonomic neuropathy; diagnostic performance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dr.Tang's research group: This group included participants with completed both the short-term HRV test and Ewing's test.
  Interventions: Other: not intervention

INTERVENTIONS:
Other: not intervention — This is a cross-sectional study for estimation of diagnostic performance.

SUMMARY:
This study aimed to evaluate the reference values for the short-term heart rate variable (HRV), estimate the performance of cardiovascular autonomic neuropathy (CAN) diagnostic tests in the absence of a gold standard, and assess CAN prevalence in our cross-sectional dataset.

DETAILED DESCRIPTION:
The CAN prevalence is rapidly growing in all populations worldwide. No document has been reported about normal reference values for CAN using this test in the Chinese population. This study aimed to evaluate the reference values for the short-term HRV in a large cross-sectional dataset, and to estimate sensitivities and specificities of CAN diagnostic tests using the Bayesian approach, in the absence of a gold standard in another independence dataset. Finally, CAN prevalence was estimated in the investigators' cross-sectional dataset. Firstly, the reference the values for the short-term HRV were calculated in the investigators' previous study (including 371 healthy subjects). This study dataset contained 88 subjects who completed both the short-term HRV test and Ewing's test. Simultaneous inferences about the population prevalence and the performance of each diagnostic test were possible using the Bayesian approach without a gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Survey participants with undiagnosed CAN, aged 30-80 years, were included in this study.

Exclusion Criteria:

* Some subjects were excluded from the study to eliminate potential confounding factors that may have influenced their CA function 11. Briefly, the exclusion criteria were as follows:

  1. history or findings of arrhythmia, and hyperthyroidism or hypothyroidism;
  2. pregnancy or lactation; and/or
  3. serious hepatic or renal dysfunctions.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with inclusion and exclusion criteria were recruited from healthy examination centres to assess cardiovascular autonomic function using both the short-term heart rate variability and Ewing's tests.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2011-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cardiovascular autonomic function evaluate by short-term heart rate variability test | participants will be measured for the duration of outpatient stay, an expected average of two days
  Both short-term heart rate variability and Ewing's test measure cardiovascular autonomic function
Cardiovascular autonomic function evaluate by Ewing's test | participants will be measured for the duration of outpatient stay, an expected average of two days
  Both short-term heart rate variability and Ewing's test measure cardiovascular autonomic function

CONTACTS AND LOCATIONS:
Overall Officials: Zihui Tang, M.D and Ph.D, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Zeng F, Tang ZH, Li Z, Yu X, Zhou L. Normative reference of short-term heart rate variability and estimation of cardiovascular autonomic neuropathy prevalence in Chinese people. J Endocrinol Invest. 2014 Apr;37(4):385-91. doi: 10.1007/s40618-013-0047-4. Epub 2014 Jan 9. PMID 24633734
- [Result] Tang ZH, Zeng F, Yu X, Zhou L. Bayesian estimation of cardiovascular autonomic neuropathy diagnostic test based on baroreflex sensitivity in the absence of a gold standard. Int J Cardiol. 2014 Feb 15;171(3):e78-80. doi: 10.1016/j.ijcard.2013.11.100. Epub 2013 Dec 6. No abstract available. PMID 24360155
- [Result] Tang ZH, Wang L, Zeng F, Li Z, Yu X, Zhang K, Zhou L. Bayesian estimation of cardiovascular autonomic neuropathy diagnostic test based on short-term heart rate variability without a gold standard. BMJ Open. 2014 Oct 6;4(9):e005096. doi: 10.1136/bmjopen-2014-005096. PMID 25287103
- [Result] Tang ZH, Zeng F, Ye K, Yu X, Zhou L. The analysis of a reference value for baroreflex sensitivity and cardiovascular autonomic neuropathy prevalence in a Chinese population. Eur J Med Res. 2014 Feb 12;19(1):8. doi: 10.1186/2047-783X-19-8. PMID 24521230